CLINICAL TRIAL: NCT07292077
Title: Frequency of Restless Legs Syndrome in Patients With Temporomandibular Joint Disorders and Its Effect on Sleep Quality
Brief Title: Restless Legs Syndrome in Temporomandibular Joint Disorders
Status: Completed | Type: Observational
Sponsor: Gulseren Demir Karakilic (Other)
Collaborators: Bozok University (Other); Gaziantep City Hospital (Other)
Responsible Party: Sponsor-Investigator, Gulseren Demir Karakilic, Assistant Professor, Principal Investigator, Bozok University
Organization: Bozok University (Other)
Other Study IDs: 140/2025
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Joint Disorders; Restless Legs Syndrome; Sleep Quality
Keywords: Temporomandibular Disorder; Restless Legs Syndrome; Sleep Quality; Mandibular Function; Quality of Life; The International Restless Legs Syndrome Study Group Diagnostic Criteria; The International Restless Legs Syndrome Study Group Criteria Severity Rating Scale; the Pittsburgh Sleep Quality Index; SF-12; Cross-sectional Study
MeSH Terms: conditions — Temporomandibular Joint Disorders; Restless Legs Syndrome; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Temporomandibular Disorder Group: This group includes adults aged 18 to 65 years who were clinically diagnosed with temporomandibular joint disorder at the otorhinolaryngology outpatient clinic of Gaziantep City Hospital, Türkiye. All participants were cognitively competent, literate, and provided written informed consent. Participants completed standardized questionnaires assessing mandibular function, symptoms of anxiety and depression, severity of restless legs syndrome, sleep quality, and health-related quality of life.
- Healthy Control Group: This group includes healthy adults without a diagnosis of temporomandibular joint disorder who were matched to the patient group for age and sex. All participants were cognitively competent, literate, and provided written informed consent. Control participants completed the same standardized questionnaires as the patient group to allow comparison of sleep quality, emotional status, and health-related quality of life between groups.

SUMMARY:
This observational, cross-sectional, descriptive study aims to evaluate the prevalence of restless legs syndrome in patients with temporomandibular joint dysfunction and to investigate its effects on sleep quality and health-related quality of life. The study will be conducted in the otolaryngology outpatient clinic of Gaziantep City Hospital, Türkiye.

Adults aged 18 to 65 years who are clinically diagnosed with temporomandibular joint dysfunction and meet the inclusion criteria will be invited to participate. An age- and sex-matched control group consisting of individuals without temporomandibular joint dysfunction will also be recruited.

All participants will undergo face-to-face structured interviews during which standardized and validated questionnaires will be administered. The study will collect sociodemographic data, clinical characteristics, and responses to validated assessment tools measuring mandibular function, anxiety and depression symptoms, restless legs syndrome, sleep quality, and health-related quality of life.

DETAILED DESCRIPTION:
This observational, cross-sectional, descriptive study aims to evaluate the prevalence of restless legs syndrome in patients with temporomandibular joint dysfunction and to investigate its effects on sleep quality and health-related quality of life. The study will be conducted in the otolaryngology outpatient clinic of Gaziantep City Hospital, Türkiye.

Adults aged 18 to 65 years who are clinically diagnosed with temporomandibular joint dysfunction and meet the inclusion criteria will be invited to participate. An age- and sex-matched control group consisting of individuals without temporomandibular joint dysfunction will also be recruited.

All participants will undergo face-to-face structured interviews during which standardized and validated questionnaires will be administered. The study will collect sociodemographic data, clinical characteristics, and responses to validated assessment tools measuring mandibular function, anxiety and depression symptoms, restless legs syndrome, sleep quality, and health-related quality of life.

The temporomandibular joint is a complex musculoskeletal structure, and temporomandibular joint dysfunction is a clinical condition involving the joint, the masticatory muscles, and surrounding tissues. Restless legs syndrome is a neurological disorder characterized by uncomfortable sensations in the legs and an uncontrollable urge to move, particularly during periods of rest or at night. Previous studies have suggested possible associations between temporomandibular joint dysfunction, bruxism, sleep disturbances, and restless legs syndrome. However, the prevalence of restless legs syndrome and its impact on sleep quality in patients with temporomandibular joint dysfunction remain insufficiently investigated.

This study is designed as an observational, cross-sectional, descriptive investigation. It will be conducted in the otolaryngology outpatient clinic of Gaziantep City Hospital and Gaziantep Dr. Ersin Arslan Training and Research Hospital. The study population will consist of adults aged 18 to 65 years who are clinically diagnosed with temporomandibular joint dysfunction, are cognitively intact, literate, and voluntarily agree to participate.

The control group will include healthy volunteers without a diagnosis of temporomandibular joint dysfunction, matched to the patient group for age and sex. Control participants will also be cognitively intact, literate, and willing to provide written informed consent.

Data Collection Tools (Final Version) Sociodemographic Questionnaire

This 25-item form records age, sex, marital status, educational level, income status, comorbidities, disease duration, and other relevant clinical characteristics.

Mandibular Functional Impairment Questionnaire

This is a 17-item questionnaire scored on a five-point Likert scale, yielding total scores ranging from 0 to 68. Higher scores indicate greater functional impairment of the mandible. The instrument evaluates patient-perceived difficulty in performing mandibular movements and daily functional tasks.

Hospital Anxiety and Depression Scale

This 14-item self-report questionnaire includes two subscales assessing anxiety and depression symptoms. Each item is scored from 0 to 3. Subscale scores range from 0 to 21, with higher scores indicating greater symptom severity.

International Restless Legs Syndrome Study Group Diagnostic Criteria

These clinical diagnostic criteria focus on the core symptoms of restless legs syndrome. Diagnosis is based on patient history and the presence of all essential diagnostic features.

International Restless Legs Syndrome Severity Scale

This 10-item rating scale evaluates symptom severity, frequency, and impact on daily life and mood. Each item is scored from 0 to 4, producing a total score between 0 and 40. Higher scores indicate greater symptom severity.

Pittsburgh Sleep Quality Index

This 24-item questionnaire assesses sleep quality over the previous month across seven components, including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Total scores range from 0 to 21, with higher scores indicating poorer sleep quality.

Short Form 12 Health Survey

This 12-item questionnaire evaluates health-related quality of life across physical and mental health domains, including physical functioning, role limitations, bodily pain, general health perception, vitality, social functioning, emotional role limitations, and mental health.

ELIGIBILITY:
Inclusion Criteria

Adults aged 18 to 65 years

For the patient group: clinical diagnosis of temporomandibular joint disorder

Cognitively intact and able to understand study procedures

Literate and able to complete self-report questionnaires

Willing to participate and provided written informed consent

Exclusion Criteria

Presence of neurological or psychiatric disorders

Cognitive impairment that interferes with questionnaire completion

Systemic diseases that may affect sleep or motor function

Current use of medications that may influence sleep or motor function

Refusal or inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study included adults aged 18 to 65 years who were recruited from the otorhinolaryngology outpatient clinic of Gaziantep City Hospital. The patient group consisted of individuals with a clinical diagnosis of temporomandibular joint disorder, while the control group comprised healthy volunteers without temporomandibular joint disorder who were matched to the patient group for age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
International Restless Legs Syndrome Study Group Diagnostic Criteria | At baseline
  This diagnostic framework defines the presence of restless legs syndrome based on standardized clinical features, including an urge to move the legs, worsening of symptoms during rest, partial or complete relief with movement, and worsening of symptoms in the evening or at night. These diagnostic criteria have been adapted for use in Turkish-speaking populations and are used to determine whether participants meet the clinical diagnosis of restless legs syndrome.
International Restless Legs Syndrome Study Group Severity Rating Scale | At baseline
  This scale consists of 10 questions assessing the severity, frequency, and impact of restless legs syndrome symptoms on daily life. Each item is scored from 0 to 4, yielding a total score ranging from 0 to 40. Higher scores indicate greater symptom severity. Severity categories are defined as mild (1-10), moderate (11-20), severe (21-30), and very severe (31-40). The Turkish version of this scale has demonstrated acceptable reliability and validity for clinical and research use.
Pittsburgh Sleep Quality Index | At baseline
  This questionnaire evaluates sleep quality over the previous month. It includes 24 items grouped into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored from 0 to 3, with a total score ranging from 0 to 21. Higher scores indicate poorer sleep quality, and a total score greater than 5 reflects poor sleep quality. The Turkish version has been shown to be valid and reliable in adult populations.

SECONDARY OUTCOMES:
Mandibular Function Impairment Questionnaire | At baseline
  This questionnaire contains 17 items assessing the individual's perceived difficulty in performing mandibular movements and daily activities such as chewing, speaking, and yawning. Each item is scored on a five-point Likert scale ranging from 0 (no difficulty) to 4 (very severe difficulty). The total score ranges from 0 to 68, with higher scores indicating greater functional impairment of the mandible. The Turkish version of this questionnaire has demonstrated satisfactory validity and reliability
Hospital Anxiety and Depression Scale | At baseline
  This self-report instrument consists of 14 items designed to assess symptoms of anxiety and depression in adults. Seven items assess anxiety symptoms and seven items assess depressive symptoms. Each item is scored from 0 to 3, producing subscale scores ranging from 0 to 21. Higher scores indicate greater symptom severity. The Turkish version has been shown to be valid and reliable in clinical populations.
12-Item Short Form Health Survey | At baseline
  This health-related quality of life questionnaire includes 12 items that assess physical and mental well-being. The instrument provides summary scores reflecting physical and mental health status, with higher scores indicating better perceived health and functioning. The Turkish version has demonstrated adequate psychometric properties for use in population-based and clinical studies

CONTACTS AND LOCATIONS:
Locations (1):
- Yozgat Bozok University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected during the study that are directly related to the primary and secondary outcomes will be made available upon reasonable request. The data will be shared exclusively for scientific and research purposes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The individual participant data and supporting documents will be available starting six months after publication of the study results and will remain accessible for a period of five years following publication.
Access Criteria: Access to the de-identified individual participant data and supporting documents will be granted to qualified researchers who submit a reasonable and scientifically valid request to the corresponding author. Requests will be reviewed by the study investigators, and access will be provided for research purposes only. Data will be shared in a secure manner through institutional data transfer or encrypted electronic communication.
URL: https://hastane.bozok.edu.tr/

REFERENCES:
- [Background] Soylu C, Kutuk B. Reliability and Validity of the Turkish Version of SF-12 Health Survey. Turk Psikiyatri Derg. 2022 Summer;33(2):108-117. doi: 10.5080/u25700. English, Turkish. PMID 35730511
- [Background] Ağargün, M.Y., Validity and reliability of Turkish version of Pittsburgh Sleep Quality Index. Türk Psikiyatri Dergisi, 1996. 7: p. 107.
- [Background] Ay, E., Huzursuz bacaklar sendromunda kullanılan uluslararası huzursuz bacaklar sendromu çalışma grubu şiddet ölçeğinin türkçe geçerlilik ve güvenilirliğinin araştırılması. 2017, Sağlık Bilimleri Enstitüsü.
- [Background] Allen RP, Picchietti DL, Garcia-Borreguero D, Ondo WG, Walters AS, Winkelman JW, Zucconi M, Ferri R, Trenkwalder C, Lee HB; International Restless Legs Syndrome Study Group. Restless legs syndrome/Willis-Ekbom disease diagnostic criteria: updated International Restless Legs Syndrome Study Group (IRLSSG) consensus criteria--history, rationale, description, and significance. Sleep Med. 2014 Aug;15(8):860-73. doi: 10.1016/j.sleep.2014.03.025. Epub 2014 May 17. PMID 25023924
- [Background] Aydemir, Ö., et al., Validity and reliability of Turkish version of hospital anxiety and depression scale. Turk Psikiyatri Derg, 1997. 8(4): p. 280-7
- [Background] Kılınç, H.E., et al., Further Validity and Reliability of Turkish Version of the Mandibular Functional Impairment Questionnaire in Patients with Temporomandibular Dysfunction. Journal of Basic and Clinical Health Sciences, 2022. 7(1): p. 214-222.